CLINICAL TRIAL: NCT04373551
Title: PrEP Demonstration Project Among Women at Risk for HIV Infection
Brief Title: WeExPAnd: PrEP Demonstration Project Among Women at Risk for HIV Infection - Preexposure Prophylaxis (PrEP)
Acronym: PrEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Mirjam-Colette Kempf, Principle Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 300003885; 1R34MH118044-01A1 (NIH)
Record Dates: First submitted 2020-04-28; First posted 2020-05-04 (Actual); Results first posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-10

CONDITIONS: HIV-infection/AIDS
Keywords: Pre exposure prophylaxis (PrEP); HIV prevention; African American women; cisgender women
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Patient: cultural adaptation of a patient-provider communication tool (Experimental): Strengthening of the PrEP care continuum by developing and testing an intervention designed to improve PrEP awareness, screening, engagement, retention, adherence, and persistence among individuals at substantial risk for HIV infection; developing and testing an intervention to reduce racial/disparities in PrEP uptake and use.
  Interventions: Behavioral: Cultural adaptation of a patient-provider communication tool

INTERVENTIONS:
Behavioral: Cultural adaptation of a patient-provider communication tool — Adaptation of a patient-provider communication tool for PrEP uptake utilized among women and their providers in a pilot pre/post-intervention design.
  Other Names: CDC PrEP tool kit

SUMMARY:
The objective of this application is to increase PrEP uptake among women vulnerable to HIV acquisition in the rural South, specifically those seeking care at Federally Qualified Healthcare Centers (FQHC) in rural Alabama.

The investigators will use a mixed-methods approach to adapt and pilot test a patient-provider communication tool from the Centers for Disease Control and Prevention (CDC) PrEP toolkit that focuses on the first three steps of the PrEP cascade (e.g., recognizing HIV risk, identifying as a PrEP candidate, and interested in PrEP) to increase PrEP uptake via referrals to local PrEP clinics.

DETAILED DESCRIPTION:
Investigators completed formative qualitative research to explore the HIV risk perceptions of African American or Black (AA) women with recent PrEP use, AA women who are candidates for PrEP, and providers and to identify preferences around patient-provider communication about HIV risk and PrEP services (Aim 1).

The investigators then systematically adapted a patient-provider communication tool to increase PrEP uptake at federally qualified health centers in Alabama, using an iterative implementation process (Aim 2A), and assessed the feasibility, acceptability, and preliminary impact of the patient-provider communication intervention on PrEP uptake among women in a pilot pre-/post-intervention design (Aim 2B).

Provider training completion rates and satisfaction with the communication tool were assessed to evaluate implementation feasibility and intervention delivery. The study systematically documented and evaluated reasons for declining PrEP referrals, incomplete referrals, failure to initiate PrEP after successful referral, and ongoing PrEP use at 3 and 12 months post-intervention.

ELIGIBILITY:
Inclusion/Exclusion Criteria

Patients

* HIV-uninfected women
* Age 18 years or older
* English speaking
* Report sexual activity or anticipate sexual activity within 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 67 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam-Colette Kempf, PhD, MPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Our data sharing plans will be discussed with our NIH program officer and based on their feedback, may be altered. Our current plans call for the results of the process and outcome evaluations collected as part of this project will be shared via professional presentations and publications, and will also be shared upon request. De-identified data will also be electronically encrypted and archived for use by others who are interested in using this data. New procedures, protocols, data collection instruments and analytic routines will be made available to interested investigators.
Supporting Information: ICF
Time Frame: Data will be available after analysis is completed.
Access Criteria: Only de-identified information will be available.

REFERENCES:
- [Result] Psaros C, Goodman GR, McDonald VW, Ott C, Blyler A, Rivas A, Shan L, Campbell M, Underwood E, Krakower D, Elopre L, Kudroff K, Sherr KH, Kempf MC. Protocol for WeExPAnd: a prospective, mixed-methods pilot demonstration study to increase access to pre-exposure prophylaxis among women vulnerable to HIV infection in the Southern USA. BMJ Open. 2023 Jun 7;13(6):e075250. doi: 10.1136/bmjopen-2023-075250. PMID 37286316

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient participants were recruited from a Federally Qualified Health Care Center (FQHC) (Site 1) and an HIV and sexually transmitted infection (STI) clinic (Site 2) in Tuscaloosa, Alabama from March 2022-June 2024. First patient participant was enrolled March 7, 2022; last participant was enrolled in June 27, 2024.
Groups:
- Patient: Cultural Adaptation of a Patient-Provider Communication Tool: The goal of the intervention is to strengthen the PrEP care continuum by developing and testing a culturally adapted patient-provider communication tool designed to improve PrEP awareness, screening, engagement, retention, adherence, and persistence among individuals at increased risk for HIV seroconversion. Specifically, the intervention aims to reduce racial and gender disparities in PrEP uptake and use.
  Each enrolled patient participant took part in a pilot study evaluating a patient-provider communication tool adapted for PrEP uptake among women and their healthcare providers, using a pre-post intervention design. Participating healthcare providers discussed PrEP with participants using the communication tool.
Period: Overall Study
Arm/Group | Patient: Cultural Adaptation of a Patient-Provider Communication Tool
Started | 67
Intervention | 53
3-month Follow-up | 53
12-month Follow-up | 48
Completed | 48
Not Completed | 19
Not completed — Lost to Follow-up | 15
Not completed — Did not collect 12-month data on participants enrolled in 2024 (at Site 2) | 4

BASELINE CHARACTERISTICS:
Groups:
- Patient: Cultural Adaptation of a Patient-Provider Communication Tool: The goal of the intervention is to strengthen the PrEP care continuum by developing and testing a culturally adapted patient-provider communication tool designed to improve PrEP awareness, screening, engagement, retention, adherence, and persistence among individuals at increased risk for HIV seroconversion. Specifically, the intervention aims to reduce racial and gender disparities in PrEP uptake and use.
  Each enrolled patient participant took part in a pilot study evaluating a patient-provider communication tool adapted for PrEP uptake among American women and their healthcare providers, using a pre-post intervention design. Participating healthcare providers discussed PrEP with participants using the communication tool.
Arm/Group | Patient: Cultural Adaptation of a Patient-Provider Communication Tool
Number analyzed (Participants) | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.6 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 67
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 65
  White | 0
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 67
Education [Count of Participants; unit: Participants]
  Some High School, No Diploma | 14
  High School Diploma/GED | 27
  Associate's/Bachelor's Degree | 23
  Graduate Degree | 3
Religion [Count of Participants; unit: Participants]
  Christian | 56
  Atheist | 1
  Other | 2
  Prefer not to answer | 8
Household Income [Count of Participants; unit: Participants]
  Less than $30,000 | 50
  $30,000 to less than $60,000 | 11
  Prefer not to answer/Unknown | 3
  Missing | 3
Primary Insurance [Count of Participants; unit: Participants]
  Medicaid/Medicare | 27
  Private Insurance (e.g., Blue Cross) | 17
  None | 19
  Other | 3
  Prefer not to answer | 1
Housing [Count of Participants; unit: Participants]
  Renting home/apartment | 42
  A friend or relative's home/apartment | 11
  Home/apartment owned by you/household member | 10
  Publicly subsidized housing | 2
  Other | 1
  Prefer not to answer | 1
Have household members living with HIV [Count of Participants; unit: Participants]
  Yes | 6
  No | 61
Relationship Status [Count of Participants; unit: Participants]
  Single/Never married | 35
  Divorced/Separated | 8
  Widowed | 1
  Prefer not to answer | 3
  Married/In a relationship | 20
Children [Count of Participants; unit: Participants]
  Yes | 43
  No | 22
  Prefer not to answer | 2
Have you heard of a daily pill that an HIV-negative person can take to prevent getting HIV? [Count of Participants; unit: Participants]
  Yes | 22
  No/Don't Know | 45
How likely would you be to take this HIV prevention pill if it were available to you for free? [Count of Participants; unit: Participants]
  Definitely would not take it | 5
  Probably would not take it | 10
  Might take it | 19
  Probably would take it | 11
  Definitely would take it | 20
  Prefer not to answer | 2
Do you plan to start taking PrEP as an HIV prevention method? [Count of Participants; unit: Participants]
  No, not thinking about it | 23
  Thinking about it; may start in the next 6 months | 21
  Thinking about it; intend to start in the next month | 10
  Yes, plan to start as soon as possible | 10
  Prefer not to answer | 3
Occupation/Income Source [Count of Participants; unit: Participants]
  Working/temporarily laid off | 37
  Disabled (permanently or temporarily) | 13
  Looking for work or unemployed | 7
  Student | 5
  Other/Prefer not to answer | 5
Have you ever taken Pre-exposure Prophylaxis (PrEP) to prevent HIV infection? [Count of Participants; unit: Participants]
  Yes | 1
  No | 66

OUTCOME MEASURES:

1. Primary Outcome: Intervention Feasibility: Enrollment Rates Among Eligible Patients Screened
Description: To determine intervention feasibility through analysis of enrollment rates (i.e., proportion of eligible patient participants who consent to participate, decline, or are lost to follow-up over the total number of eligible patient participants screened) and reasons for declining enrollment.
Time Frame: Throughout recruitment period (approximately 24 months)
Population: HIV-uninfected women aged 18 years or older who are English-speaking and report sexual activity or anticipate sexual activity within 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patient: Cultural Adaptation of a Patient-Provider Communication Tool
Number analyzed (Participants) | 215
Participants
  Enrolled | 67
  Declined: No interest in research | 60
  Declined: Does not feel at risk for HIV | 27
  Declined: No time | 37
  Declined: New medication hesitancy | 2
  Declined: Other - already on PrEP | 2
  Declined: Multiple reasons | 5
  Declined: No reason provided | 3
  Lost to follow-up | 12

2. Primary Outcome: Intervention Feasibility: Intervention Completion Rates Among Enrolled Patients
Description: To determine intervention feasibility through the analysis of intervention completion rates (i.e., proportion of enrolled patient participants who completed the intervention) and reasons for incomplete intervention
Time Frame: Throughout recruitment period (approximately 24 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Patient: Cultural Adaptation of a Patient-Provider Communication Tool
Number analyzed (Participants) | 67
Participants
  Complete intervention | 53
  Incomplete intervention (i.e., lost to follow-up) | 14

3. Primary Outcome: Intervention Feasibility: 3-month Follow-up Completion Rates Among Patients With Completed Intervention
Description: To determine intervention feasibility through the analysis of 3-month follow-up completion rates (i.e., proportion of enrolled patient participants with complete interventions with complete 3-month follow-up data)
Time Frame: Throughout recruitment and follow-up period (approximately 24 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Patient: Cultural Adaptation of a Patient-Provider Communication Tool
Number analyzed (Participants) | 53
Participants | 53

4. Primary Outcome: Intervention Feasibility: PrEP Referral Acceptance Among Patients With Completed Intervention
Description: To determine intervention feasibility through the analysis of PrEP referral acceptance rates (i.e., proportion accepting PrEP referral among those offered) and reasons for declining a referral
Time Frame: Throughout recruitment period and follow-up period (approximately 24 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Patient: Cultural Adaptation of a Patient-Provider Communication Tool
Number analyzed (Participants) | 53
Participants
  Accepted PrEP Referral | 18
  Declined PrEP: Low perceived HIV risk | 12
  Declined PrEP: New medication hesitancy | 5
  Declined PrEP: Need for more information/consideration time | 5
  Declined PrEP: Logistical/timing concerns | 1
  Declined PrEP: Delayed PrEP referral acceptance after intervention | 1
  Declined PrEP: Reason unknown | 11

5. Primary Outcome: Intervention Acceptability: Client Satisfaction Among Patients With Completed Intervention
Description: To determine intervention acceptability using the Client Satisfaction Questionnaire (CSQ-8), an 8-item instrument that measures patient participants' perceived value of the intervention. The CSQ-8 generates a total score by summing individual item responses, with possible scores ranging from 8 to 32, where higher scores reflect greater treatment satisfaction.
Time Frame: On intervention day, directly after intervention delivery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient: Cultural Adaptation of a Patient-Provider Communication Tool
Number analyzed (Participants) | 53
score on a scale | 30.45 (1.78)

6. Primary Outcome: Preliminary Effectiveness: PrEP Uptake Among Eligible Patients Post-Intervention
Description: To determine preliminary effectiveness through PrEP uptake (i.e., proportion of patient participants who initiated PrEP (i.e., got PrEP prescription) over the number of eligible patients referred to PrEP) in the participating clinic post-intervention.
Time Frame: Enrollment to 3 months post-intervention
Population: The overall number of participants analyzed for this outcome measure includes the number of eligible patients referred to PrEP at our primary partnering clinic site (i.e., Site 1) after the intervention as part of the study (n = 17). Data from our secondary clinic site (Site 2) were excluded from the pre-post comparison due to insufficient sample size.
Measure: Number (95% Confidence Interval); unit: percentage of patients initiating PrEP
Arm/Group | Patient: Cultural Adaptation of a Patient-Provider Communication Tool
Number analyzed (Participants) | 17
percentage of patients initiating PrEP | 41.18 [21.56 to 64.05]

7. Secondary Outcome: PrEP Medication Adherence: Self-Reported PrEP Prescription Regimen Adherence Among Patients Who Initiated Oral PrEP at Both Site 1 and Site 2
Description: To determine PrEP medication regimen adherence, patient participants completed an adherence questionnaire using a 6-point Likert scale to self-report their perceived ability to take their PrEP medication as prescribed over the last 4 weeks. The scale ranged from excellent to very poor.
Time Frame: 3-month Follow-up
Population: HIV-uninfected women aged 18 years or older who are English-speaking and report sexual activity or anticipate sexual activity within 6 months; specifically, the Number of Participants Analyzed for this measure is a subset of the total number of participants who completed 3-month follow-up (n=53) and both accepted a PrEP referral and initiated oral PrEP medication after the intervention at both Site 1 and Site 2 (n=7).
Measure: Count of Participants; unit: Participants
Arm/Group | Patient: Cultural Adaptation of a Patient-Provider Communication Tool
Number analyzed (Participants) | 7
Participants
  Excellent | 1
  Very Good | 2
  Good | 2
  Fair | 2
  Poor | 0
  Very Poor | 0

8. Secondary Outcome: PrEP Medication Adherence: Self-Reported PrEP Prescription Dosage Adherence Among Participants Who Initiated Oral PrEP at Both Site 1 and Site 2
Description: To determine PrEP medication dosage adherence, patients completed an adherence questionnaire to self-report the percentage of PrEP medication they have taken in the last 4 weeks.
Time Frame: 3-Month Follow-up
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of medication taken
Arm/Group | Patient: Cultural Adaptation of a Patient-Provider Communication Tool
Number analyzed (Participants) | 7
percentage of medication taken | 72.14 (22.33)

9. Secondary Outcome: PrEP Clinic Visit Adherence at 3-months: Percentage of Scheduled PrEP Visits Attended Among Patients Who Initiated Oral or Injection PrEP at Both Site 1 and Site 2
Description: To determine PrEP clinic visit adherence, we calculated the average percentage of PrEP visits attended among patient participants who initiate PrEP, compared to the number of PrEP visits scheduled. Visit data was extracted from patients' electronic medical records.
Time Frame: From enrollment to 3-months post-enrollment
Population: HIV-uninfected women aged 18 years or older who are English-speaking and report sexual activity or anticipate sexual activity within 6 months; specifically, the Number of Participants Analyzed for this measure is a subset of the total number of participants who completed 3-month follow-up (n=53) and both accepted a PrEP referral and initiated oral or injection PrEP medication after the intervention (n=8) at both Site 1 and Site 2.
Measure: Mean (Standard Deviation); unit: percentage of PrEP visits attended
Arm/Group | Patient: Cultural Adaptation of a Patient-Provider Communication Tool
Number analyzed (Participants) | 8
percentage of PrEP visits attended | 95.83 (11.78)

10. Secondary Outcome: PrEP Clinic Visit Adherence at 12-months: Percentage of Scheduled PrEP Visits Attended Among Patients Who Initiated Oral or Injection PrEP at Site 1
Description: To determine PrEP clinic visit adherence, we calculated the average percentage of PrEP visits attended among patient participants who initiated PrEP, compared to the number of PrEP visits scheduled. Visit data was extracted from patients' electronic medical records.
Time Frame: From enrollment to 12-months post-enrollment
Population: HIV-uninfected women aged 18 years or older who are English-speaking and report sexual activity or anticipate sexual activity within 6 months; specifically, the Number of Participants Analyzed for this measure is a subset of the total number of participants who completed 12-month follow-up (n=48) and both accepted a PrEP referral and initiated oral or injection PrEP medication after the intervention at Site 1 (n=7). No 12-month data was collected from Site 2.
Measure: Mean (Standard Deviation); unit: percentage of PrEP visits attended
Arm/Group | Patient: Cultural Adaptation of a Patient-Provider Communication Tool
Number analyzed (Participants) | 7
percentage of PrEP visits attended | 85.24 (20.35)

ADVERSE EVENTS:
Time Frame: 2 years, 3 months
Description: Adverse events are harmful occurrences to study participants, either study-related or non-study related.
  Study participation reflected a unique opportunity to provide referrals for social services as we collected data on depressive symptoms and intimate partner violence. Any participant who endorsed significant symptoms on either of these measures (or a participant who spontaneously reported these problems) was provided with a referral for services from the partnering clinic.
Groups:
- Cultural Adaptation of a Client-Provider Communication Tool: The goal of the intervention is to strengthen the PrEP care continuum by developing and testing a culturally adapted client-provider communication tool designed to improve PrEP awareness, screening, engagement, retention, adherence, and persistence among individuals at increased risk for HIV seroconversion. Specifically, the intervention aims to reduce racial and gender disparities in PrEP uptake and use.
  Each enrolled participant took part in a pilot study evaluating the client-provider communication tool adapted for PrEP uptake among Black or African American cis-gender women and their healthcare providers in a pre-post intervention design. Eligibility criteria was expanded to include women of any race/ethnicity. Participating healthcare providers discussed PrEP with participants using the communication tool.
Arm/Group | Cultural Adaptation of a Client-Provider Communication Tool
All-Cause Mortality (participants affected / at risk) | 0/67
Serious Adverse Events (participants affected / at risk) | 0/67
Other Adverse Events (participants affected / at risk) | 0/67

LIMITATIONS AND CAVEATS:
Target enrollment was not met due to recruitment challenges, which limited the study's statistical power to detect intervention effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-17): https://cdn.clinicaltrials.gov/large-docs/51/NCT04373551/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-02): https://cdn.clinicaltrials.gov/large-docs/51/NCT04373551/ICF_001.pdf